CLINICAL TRIAL: NCT04458792
Title: Development of a Monocentric and Prospective Clinical and Biological Database in Sarcoma
Brief Title: Establishment of a Prospective Clinical-biological Database
Acronym: BCBSarcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-BDD 2016/03
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma
Keywords: biological specimen banks; radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Biological collection (Experimental): For all the patients include in the study :
  * Paraffin tissue samples collected during surgery (neoplasic tissue and normal tissue)
  * MDM2 project : Blood samples collected at different times : Before the surgery, and 1 month after the surgery
  * circulant DNA project : Blood samples collected at different times : Before the surgery, and 1 month after the surgery
  * radiotherapy toxicity : Blood samples collected before the radiotherapy
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Paraffin tissue samples; Other: blood sample

INTERVENTIONS:
Other: Paraffin tissue samples — Paraffin tissue samples collected during surgery (neoplasic tissue and normal tissue
Other: blood sample — MDM2 project : Blood samples collected at different times : Before the surgery, and 1 month after the surgery circulant DNA project : Blood samples collected at different times : Before the surgery, and 1 month after the surgery radiotherapy toxicity : Blood samples collected before the radiotherapy

SUMMARY:
A Clinical and Biological Database will provide to the scientific community a collection of blood and tissues with clinical data to improve knowledge about cancer and help to develope new cancer treatments. This database is specific to Sarcoma

DETAILED DESCRIPTION:
Liposarcomas (LPS) are soft tissue tumours of mesenchymal origin. The most common histological subtypes, represented by well differenciated Lipsarcomas (WD-LPS) and dedifferenciated (DD-LPS), are characterized by the quasi-systematic amplification of the q13-15 of chromosome 12 containing the Mdm2 gene.

The systematic amplification of the Mdm2 gene is such that it is used clinically to distinguish WD/DD-LPS from other types of sarcomas. These observations raise key questions about the high selection pressure that leads to the almost systematic amplification of Mdm2 during the development of these LPS.

Mdm2 is an oncoprotein whose roles in p53 tumour suppressor degradation are broadly described. However, the different inhibitors targeting this interaction were disappointing in clinical trials.

Recently a team from the U1194 INSERM unit of the IRCM which collaborates in this project showed by a pan-genomics analysis, that Mdm2 is recruited to chromatin within a multiproteic complex having as target a transcriptional program involved in the metabolism and in particular in the biosynthesis of the serin.

This clinical-biological basis will allow the continuation of this research project on liposarcomas and the development of new research projects on other histological types of sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* men or women > 18 years
* Patient treated by surgery for : a primitive sarcoma and/or local relapse sarcoma and/or metastatic localisation of sarcoma
* patient accepted blood sample
* patient treated by radiotherapy before or after the surgery
* Patient signed informed consent

Exclusion Criteria:

* Patient not affiliated to french Social Protection system
* Patient under guardianship
* Patient unable to understand or comply with study instructions or requirements for psychological, family, social or geographical reasons
* Pregnancy and/or feeding
* Patient take care in an Emergency Situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Establishment a clinical and biological database will provide to the scientific community a collection of blood and tissues with clinical data to improve knowledge about sarcoma | Until the study completion : 5 years
  number of collection of tissue samples (tumour tissue and healthy tissue) in patients operated on a sarcoma associated with clinical data.
Establishment a clinical and biological database will provide to the scientific community a collection of blood and tissues with clinical data to improve knowledge about sarcoma | Until the study completion : 5 years
  Number of collection of blood in patients operated on a sarcoma associated with clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: FIRMIN Nelly, MD, Study Chair — Institut régional du Cancer Montpellier
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Peoc'h M, Istier L, Chalabreysse P, Muller C, Alberti L, Bringuier PP, Scoazec JY, Schott AM, Bergeron C, Cellier D, Blay JY, Ray-Coquard I. Incidence of sarcoma histotypes and molecular subtypes in a prospective epidemiological study with central pathology review and molecular testing. PLoS One. 2011;6(8):e20294. doi: 10.1371/journal.pone.0020294. Epub 2011 Aug 3. PMID 21826194
- [Result] Mastrangelo G, Coindre JM, Ducimetiere F, Dei Tos AP, Fadda E, Blay JY, Buja A, Fedeli U, Cegolon L, Frasson A, Ranchere-Vince D, Montesco C, Ray-Coquard I, Rossi CR. Incidence of soft tissue sarcoma and beyond: a population-based prospective study in 3 European regions. Cancer. 2012 Nov 1;118(21):5339-48. doi: 10.1002/cncr.27555. Epub 2012 Apr 19. PMID 22517534
- [Result] Crago AM, Singer S. Clinical and molecular approaches to well differentiated and dedifferentiated liposarcoma. Curr Opin Oncol. 2011 Jul;23(4):373-8. doi: 10.1097/CCO.0b013e32834796e6. PMID 21552124
- [Result] Lokka S, Scheel AH, Dango S, Schmitz K, Hesterberg R, Ruschoff J, Schildhaus HU. Challenging dedifferentiated liposarcoma identified by MDM2-amplification, a report of two cases. BMC Clin Pathol. 2014 Jul 28;14:36. doi: 10.1186/1472-6890-14-36. eCollection 2014. PMID 25126005
- [Result] Marine JC, Lozano G. Mdm2-mediated ubiquitylation: p53 and beyond. Cell Death Differ. 2010 Jan;17(1):93-102. doi: 10.1038/cdd.2009.68. PMID 19498444
- [Result] Ray-Coquard I, Blay JY, Italiano A, Le Cesne A, Penel N, Zhi J, Heil F, Rueger R, Graves B, Ding M, Geho D, Middleton SA, Vassilev LT, Nichols GL, Bui BN. Effect of the MDM2 antagonist RG7112 on the P53 pathway in patients with MDM2-amplified, well-differentiated or dedifferentiated liposarcoma: an exploratory proof-of-mechanism study. Lancet Oncol. 2012 Nov;13(11):1133-40. doi: 10.1016/S1470-2045(12)70474-6. Epub 2012 Oct 17. PMID 23084521